CLINICAL TRIAL: NCT04953403
Title: Evaluation of Physical Activity of Patients Admitted to Addiction Service
Acronym: ACTP-ADDICT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0374
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Alcoholism
Keywords: Psychoactive substances consumption; Physical activity; Alcohol withdrawal; Dependence level; Drug users
MeSH Terms: conditions — Alcoholism; Motor Activity; Drug Misuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Addiction is a public health issue that affects nearly 30% of French people according to INSEE. For several years now, the investigators have known that sport is a real help in the fight against addictions, with recent medical authorization to prescribe physical activities. A study from August 2016 claims that regular physical activity may offset the harmful effects of alcohol. (1) Based on the answers given by 36,370 Britons between 1994 and 2006, the researchers showed the existence of a link between the practice of 150 minutes of physical activity per week and the decrease in deaths linked to consumption. alcohol. These results, compared to 18 other studies (2), reveal the benefits of physical activity in the management of addictions. But what about current practice and addictions and sports practice in general ?

ELIGIBILITY:
Inclusion criteria:

- Any patient entering the addictology service for a reason related to addiction (withdrawal, VMI, etc.) at the CHU de St Eloi between January 01, 2020 and May 31, 2020 aged at least 18 years old

Exclusion criteria:

* Patient whose hospitalization is not related to addictology (accommodation, medical examination, etc.)
* Minor patient (age <18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient entering the addictology service for a reason related to addiction (withdrawal, VMI, etc.) at the CHU de St Eloi between January 01, 2020 and May 31, 2020 aged at least 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Assess the relationship between the level of physical activity of patients hospitalized for drug addiction withdrawal | 5 months
  Assess the relationship between the level of physical activity of patients hospitalized for drug addiction withdrawal
Assess the relationship between the level of physical activity of patients hospitalized for dependence on alcohol and tobacco | 5 months
  Assess the relationship between the level of physical activity of patients hospitalized for dependence on alcohol and tobacco
level of physical activity of patients | 5 months
  level of physical activity of patients
The relationship between the level of physical activity before the onset of dependence | 5 months
  The relationship between the level of physical activity before the onset of dependence

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Donnadieu-Rigole, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC